CLINICAL TRIAL: NCT06063525
Title: Biological Implications of the Overlapping Phenomenon Between Childhood Schizophrenia and Autism Spectrum Disorders-Heterogeneity Approach Rather Than Diagnostic Boundary
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201412165RINB
Record Dates: First submitted 2023-05-04; First posted 2023-10-02 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-01

CONDITIONS: Schizophrenia; Autism Spectrum Disorder
MeSH Terms: conditions — Schizophrenia; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- childhood onset schizophrenia (COS): diagnosis of schizophrenia under the age of 13 years.
  Interventions: Other: Structural anatomy
- schizophrenia (SZ): patients with schizophrenia with and age of onset later than 13 years
  Interventions: Other: Structural anatomy
- autism spectrum disorder (ASD): dual diagnosis of schizophrenia and ASD, including SZ with ASD, COS with ASD
  Interventions: Other: Structural anatomy

INTERVENTIONS:
Other: Structural anatomy — images acquired with 3T MRI system with 32 channel head coil

SUMMARY:
Complex diseases such as schizophrenia and autism are heterogeneous in clinical presentation and etiology. This high heterogeneity constitutes the challenges for the clinical diagnosis and etiological research, resulting in that the majority of research findings cannot be replicated in the independent samples. For the high comorbid rate between the diagnoses of schizophrenia and autism spectrum disorders (ASD), and the shared neurocognitive deficits, genetic risks, and biological markers between the two disorders, a heterogeneity approach may probably be more promising than to arbitrarily split the two diagnostic categories apart or lump them together for etiological research. In schizophrenia, patients with a very early onset of disease and with preceding neurodevelopmental conditions may imply a different underlying etiology from those with typical onset and without neurodevelopmental conditions. Echoing the evidence that in early onset Parkinson's disease, PARK2 (encoding parkin protein) mutations are successfully reported to be as frequent as 49% with an autosomal-recessive mode of inheritance , representing a specific disease entity of Parkinson's disease. Therefore, it is critical to characterize the clinical phenotypes for this subpopulation of very early onset patients, including their clinical manifestation, disease course, and treatment response, as well as early developmental history and morphological characteristics. These may establish an important base for investigating the etiology and providing adequate clinical care for the heterogeneous syndrome of schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* SZ group: schizophrenia onset earlier than 12 years old
* COS group: schizophrenia onset later than 12 years old
* ASD group: diagnosed with autism spectrum disorder without schizophrenia
* Dual group: diagnosed with ASD and SZ

Exclusion Criteria:

* congenital disease
* major physical diseases
* neurodegenerative disorder
* chromosomal aberration

Ages: 15 Years to 59 Years | Sex: All
Age Groups: Child, Adult
Study Population: as mentioned earlier, patients with schizophrenia and/or autism spectrum disorder
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2015-02-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale PANSS | 3 years
  33 item scale composed of 7 positive scale, 7 negative scale, 16 general psychopathology, and 3 aggression risk profile. Range from 0 to 7, higher the score, more severe the symptoms are.
Autism Diagnostic Observation Schedule | 3 years.
  interview with subjects. range from 0 to 8, higher the score, worse the autistic symptoms.
Physical anomalies and craniofacial features | 3 years
  41 qualitative items were used to examine the presence or absence of morphological anomalies and magnitude of anomalies. Minor physical anomalies were rated from 0 to 83, higher the score, greater the anomalies.
Brain structural anatomy with MRI scan | 3 years
  3 Tesla MRI with a 32-channel head coil was used to collect brain imaging of cortical thickness, cortical volume, white matter volume, gyrification. The MRI structural images will be analyzed using FreeSurfer image analysis suite.